CLINICAL TRIAL: NCT06667947
Title: Effect of Caudal vs. Penile Block on the Incidence of Hypospadias Complications Following Primary Repairs: A Randomized Controlled Trial
Brief Title: Effect of Caudal vs. Penile Block on the Incidence of Hypospadias Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fikret Salık, Associate professor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Dicle University
Record Dates: First submitted 2024-03-08; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Complication of Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Caudal Block
  Interventions: Procedure: caudal block
- Group 2 (Active Comparator): Penile Block
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: caudal block — For the caudal block, a caudal needle was used by the same anesthesiologist after the patients were placed in the left lateral decubitus position.
  Other Names: penile block

SUMMARY:
Hypospadias is one of the most common congenital malformations in male babies, affecting approximately 1 in every 200-300 live male births. This condition is characterized by an abnormal location of the urethral meatus, located on the ventral side of the penis, anywhere from the glans to the perineum.

Treatment of hypospadias is primarily surgical and aims at functional and cosmetic correction. However, surgery is often complex and can be associated with a significant risk of complications, such as fistula formation, wound dehiscence, urethral stricture, and dissatisfaction with cosmetic results. The search for optimal surgical techniques and postoperative management strategies that can reduce these complications continues.

Postoperative pain after penile surgery can cause agitation and anxiety in children, which can also lead to stress and tension in parents. In addition to ensuring the comfort of both children and parents, pain control reduces complications in the postoperative period and accelerates recovery. Different techniques such as local anesthesia, sedoanalgesia, general anesthesia or regional anesthesia are used in penile surgery. Caudal nerve block, a regional anesthesia technique, is widely used in pediatric infraumbilical surgeries, its anesthetic safety and effectiveness have been proven in recent years, and caudal block is generally applied safely to provide postoperative analgesia in these patients. These block applications reduce the need for analgesic and anesthetic drugs and prolong the pain-free period. At the same time, this method is easy and safe to apply. However, some anesthetic complications of caudal block have been reported in previous studies6. It has also been suggested that the use of caudal nerve block is a potential risk factor contributing to surgical complications in hypospadias surgeries. This was first reported by Kundra and his team in 2012. In the study, they noted that the fistula rate increased to 19.2% in patients receiving caudal nerve block compared to a 0% fistula rate in those receiving penile block during one-stage hypospadias repair. Since the initial findings of Kundra and his team, the use of caudal anesthesia during hypospadias repair has been a subject of ongoing debate.

Caudal nerve block, a regional anesthesia technique, is widely used in pediatric infraumbilical surgeries, and its safety and effectiveness as an anesthetic are well established. The purpose of this study was to evaluate the potential effect of caudal nerve block anesthesia on postoperative surgical outcomes in male patients aged 6-48 months undergoing hypospadias repair

ELIGIBILITY:
Inclusion Criteria:

* hypospadias

Exclusion Criteria:

* the patients who alder than 48 month

Ages: 6 Months to 48 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
complication rate | 01.07.2023-01.03.2024
  Surgery-related complications such as wound dehiscence, fistula formation, and urethral stenosis due to the surgical procedure will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle University, Sur, Di̇yarbakir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ı will individual participant data (IPD) available to other researchers.